CLINICAL TRIAL: NCT00578292
Title: Pilot Study of Allogeneic Stem Cell Transplantation From Unrelated Donors for Patients With Severe Homozygous Beta 0/+ Thalassemia or Severe Variants of Beta 0/+ Thalassemia
Brief Title: Allogeneic Stem Cell Transplantation, Severe Homzygous 0/+Thalassemia or Sever Variants of Beta 0/+ Thalassemia, THALLO
Acronym: THALLO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stem cell transplant was determined SOC for this disease (study is not relevant)
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Tami D. John, Assistant Professor, Hematology/Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THALLO (H-14539); H-14539 (Other: Baylor College of Medicine IRB)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Thalassemia
Keywords: transfusion-dependent; homozygous b0/+-thalassemia; severe variants of b0/+-thalassemia; transfusion; iron chelating agents; severe; transfusion-dependent homozygous
MeSH Terms: conditions — Thalassemia; Lymphoma, Follicular | interventions — Busulfan; fludarabine; fludarabine phosphate; Alemtuzumab; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bone Marrow or Stem Cell Infusion (Experimental): Mesna, Cyclophosphamide, Busulfan, Fludarabine, Campath 1H
  Bone Marrow or Stem Cell infusion with pre-meds to take place on Day 0.
  Bone marrow dose/stem cell dose: To ensure the probability for bone marrow engraftment, 4 x 10e8 nucleated cells/kg patient weight or 5 x 10e6/kg of CD34+ cells/kg patient weight if the product is mobilized peripheral blood, will be the target to be obtained from the unrelated donor.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Campath 1H; Drug: Cyclophosphamide; Drug: MESNA

INTERVENTIONS:
Drug: Busulfan — 4.0 mg/kg/day divided into four doses daily for four days; total dose = 16 mg/kg
  Days -9 through -6
  Other Names: Myleran
Drug: Fludarabine — 30mg/m2 Day -5 through Day -2
  Other Names: Fludara
Drug: Campath 1H — Per institutional guidelines Days -5 through -2
  Other Names: Alemtuzumab
Drug: Cyclophosphamide — 50 mg/kg Days -5 through -2
  Other Names: Cytoxan
Drug: MESNA — 10 mg/kg x 5 Days -5 through -2
  Other Names: Mesnex

SUMMARY:
Patients have severe beta-thalassemia or one of the thalassemia variants. Thalassemia is a hereditary disease in which the bone marrow produces abnormal red blood cells that have a shorter life span than normal red blood cells. Because of that, the patient has chronically low red blood cell numbers (anemia) and need regular blood transfusions to help the patient feel better and to help prevent damage to important organs such as the heart. The following treatments are currently available to patients: lifelong blood transfusions and drugs that help remove iron from the body, and long-term antibiotics to prevent infections. These treatments are difficult for patients to take, and do not stop the effects of the disease.

Currently, the only treatment that may cure thalassemia is bone marrow or blood stem cell transplantation. Special blood or bone marrow cells from a healthy person might allow the bone marrow to create healthy cells, which will replace the abnormal red blood cells of thalassemia. There is a lot of experience using special blood or bone marrow cells from a healthy brother or sister who is the same HLA (immune) type. For patients who do not have such a donor in the family, an unrelated volunteer donor can be used. It is important for the patient to realize that this kind of transplant can have more problems than a transplant from a brother or sister.

Because we do not know the long-term effects of this treatment and because this type of transplant has not been used often for people with thalassemia, this is a research study. We hope, but cannot promise, that the transplanted marrow/stem cells will produce healthy cells and the patient will no longer have severe thalassemia.

DETAILED DESCRIPTION:
To be treated on this study, we will test the blood to check for viruses, including HIV (the virus that causes AIDS). If the HIV test is positive, a transplant cannot be done because it would be too dangerous for the patient. Secondly, we will do a liver biopsy to determine if the liver has been damaged (which can happen from iron overload that develops after many transfusions). Too much liver damage could mean that the patient will have a higher risk to develop problems with the transplant.

To participate in this study, the patients also need to have a central line (a thin plastic catheter or tube that is placed during surgery into one of the large veins in the neck or chest). Central lines are used to give intravenous medications (go directly into the vein) or to take blood samples without the patient having to endure frequent needle sticks. Before the treatment starts, we will remove a small amount of the bone marrow (back-up bone marrow) and store it. The reason for this is that if the donors bone marrow or blood stem cells do not grow properly after the transplant and the patients blood counts stay low, we can put the patients own bone marrow cells back into their body. This will help the blood counts to recover, but this means that the patient will also have thalassemia again.

To prepare the body for the transplant, the patients own blood forming system has to be destroyed and their immune system has to be weakened. To do this, they will be given high dose chemotherapy and medications that weaken their immune system (also called a conditioning treatment) for 9 days before the transplant. The main chemotherapy drugs used in the conditioning treatment are: cyclophosphamide, fludarabine and busulfan. The chemotherapy treatment will last 9 days. The patient will be admitted 10 days before the transplant to start a medicine to prevent seizures before they receive the first dose of busulfan since one of the side effects of busulfan is risk of seizures. First the patient will be given a drug called busulfan through the central line every 6 hours starting 9 days before transplant (called Day -9) until 6 days before transplant (called Day -6). Starting one day after receiving the last busulfan dose (Day -5), they will receive cyclophosphamide, fludarabine and Campath IH, which will all be given through the central line once a day for the next four days. Campath IH is a special type of protein called an antibody that works against certain types of blood cells. Also on Day -5, we will add a drug called MESNA. MESNA is used to decrease the side-effects caused by cyclophosphamide.

One day after the chemotherapy treatment is finished (Say -1) the patient will have a day to rest. On Say 0, the patient will receive the bone marrow/stem cells from the donor. Once in the bloodstream, the cells will go to the bone marrow and should begin to grow. To help prevent a problem call graft-versus-host disease (GVHD), the patient will receive a small dose of methotrexate on four different days after transplant. Another drug to help prevent GVHD, tacrolimus, will be started 2 days (Day -2) before the transplant and continued for approximately one year after the transplant. To tell whether the transplant has "taken" or "engrafted", we will take samples of blood two to three weeks after the transplant.

The patient will need to be in the hospital for at least 4 weeks after the transplant to make sure the transplant has engrafted. To find out how much the treatment has helped them and how much it might help other patients, we will do several routine lung, kidney, and liver tests, including liver biopsies, after the bone marrow/stem cell transplant. Additionally, we will be looking at the immune function. To do this, we will take 30 mL (2 tablespoonfuls) of blood every three months for the first year after transplant and then every 6 months during the second year after transplant. When possible, the blood that is taken will be taken through an existing IV line. However, at times drawing the blood will require another stick with a needle. The total amount of blood to be taken will not exceed 12 tablespoonfuls.

Because bone marrow/stem cell transplant from an unrelated volunteer donor is a new therapy for severe thalassemia and because problems may happen months afterward, the patient will need to have exams and blood tests done every few months during the first and second year following transplantation.

The patient may still need to use iron removing agents for some time after transplant or undergo blood-letting to get rid of the excess iron in the body. During that time, we will monitor the amount of iron in the body. Looking at the iron stored in the liver can most accurately tell us how much excess iron the patient has in the body. We will do liver biopsies once or twice per year if the patient is receiving iron chelation treatment after the transplant.

ELIGIBILITY:
Inclusion Criteria:

Patients with documented diagnosis of severe (transfusion-dependent) homozygous b0/+-thalassemia or severe variants of b0/+-thalassemia requiring chronic transfusion therapy and iron chelating agents, who fulfill the following conditions:

1. Patient does not have an HLA genotype-identical donor available and has a 5/6 or 6/6 matched unrelated donor, or a 5/6 matched related donor available.
2. Must be between 1 and 16 yrs of age (all Pesaro risk groups).
3. Patients older than 17 yrs of age must be in Pesaro Risk Class 2 or lower (see Appendix B).
4. Women of childbearing potential must have a negative pregnancy test.
5. Documentation of compliance with iron chelation, absence or presence of hepatomegaly, and presence or absence of hepatic fibrosis prior to transplant (criteria for the Pesaro Risk Classification). This information will be obtained by history, physical exam and interpretation of liver biopsy results.
6. Documentation of awareness of alternative treatment options.

Exclusion Criteria:

1. Biopsy-proven chronic active hepatitis or fibrosis with portal bridging.
2. Has previous history of malignancies.
3. Creatinine clearance < 35 mL/min/1.73 M2.
4. Severe cardiac dysfunction defined as shortening fraction < 25%.
5. HIV infection.
6. Inadequate intellectual capacity to give informed consent (in the case of minors, this criteria must be fulfilled by the legal guardian).
7. Be pregnant, lactating or unwilling to use appropriate birth control.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2004-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tami John, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital; Tami John, MD, Study Director — Baylor College of Medicine - Texas Children's Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow or Stem Cell Infusion: Mesna, Cyclophosphamide, Busulfan, Fludarabine, Campath 1H
  Bone Marrow or Stem Cell infusion with pre-meds to take place on Day 0.
  Bone marrow dose/stem cell dose: To ensure the probability for bone marrow engraftment, 4 x 10e8 nucleated cells/kg patient weight or 5 x 10e6/kg of CD34+ cells/kg patient weight if the product is mobilized peripheral blood, will be the target to be obtained from the unrelated donor.
  Busulfan: 4.0 mg/kg/day divided into four doses daily for four days; total dose = 16 mg/kg
  Days -9 through -6
  Fludarabine: 30mg/m2 Day -5 through Day -2
  Campath 1H: Per institutional guidelines Days -5 through -2
  Cyclophosphamide: 50 mg/kg Days -5 through -2
  MESNA: 10 mg/kg x 5 Days -5 through -2
Period: Overall Study
Arm/Group | Bone Marrow or Stem Cell Infusion
Started | 10
Completed | 7
Not Completed | 3
Not completed — Death | 1
Not completed — Graft failure | 2

BASELINE CHARACTERISTICS:
Population: Participants received allogeneic hematopoietic stem cell transplantation (SCT) from unrelated donors.
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 6 [2 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Rate After Transplant
Description: Engraftment is defined as an absolute neutrophil count (ANC) >500/microL x 3 days.
Time Frame: up to 30 days
Population: The analysis included all participants who underwent allogeneic hematopoietic stem cell transplantation (SCT) from unrelated donors.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 10
proportion of participants | 1 [0.69 to 1]

2. Primary Outcome: Number of Participants With Stable Mixed Hematopoietic Chimerism (HC)
Description: Stable hematopoietic chimerism is defined as having 50-99 percent of donor cells.
Time Frame: 1 year post-transplant
Population: The analysis included all participants who underwent allogeneic hematopoietic stem cell transplantation (SCT) from unrelated donors and had mixed chimerism (MC). Six participants were not evaluable at the time point of assessment for this outcome measure due to death or graft failure or full donor.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 4
Participants | 3

3. Primary Outcome: Number of Participants With Transient Mixed Hematopoietic Chimerism (HC)
Description: Transient mixed hematopoietic chimerism is defined as any mixed chimerism return to 100 percent donor.
Time Frame: 1 year post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 4
Participants | 0

4. Primary Outcome: Number of Participants With Infectious Complications
Description: All AEs and SAEs (including infections) will be collected for evaluation of infectious complications.
Time Frame: up to day 100
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 10
Participants | 7

5. Primary Outcome: Hematopoietic Reconstitution
Description: Hematopoietic: defined as transfusion independence.
Time Frame: 1 year post-transplant
Population: The analysis included all participants who underwent allogeneic hematopoietic stem cell transplantation (SCT) and were evaluable for the outcome measure. Two participants were not evaluated at the time point of assessment for this outcome measure due to death or graft failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 8
Participants | 7

6. Primary Outcome: Immune Reconstitution
Description: Immune reconstitution: defined as absolute lymphocyte count (ALC) >1000x10e3/microL
Time Frame: 1 year post-transplant
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 8
Participants | 8

7. Primary Outcome: Number of Participants With ACUTE GVHD
Description: Acute GVHD is graded by the method of Przepiorka D. et al, which evaluates skin involvement, lower and upper GI, and liver function (bilirubin), each being graded in stages from 0 to 4, where 0 means no acute GVHD, and 4 is the highest stage of acute GVHD
Time Frame: Assessed weekly from Day 0 to day 100
Population: The analysis included all participants who underwent allogeneic hematopoietic stem cell transplantation (SCT) and were evaluable for acute GVHD. A participant is evaluable for acute GVHD if he/she engrafted and either completed 100 days observation after transplant or experienced acute GVHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 10
Participants
  Grade 0 | 4
  Grade I | 4
  Grade II-IV | 2

8. Primary Outcome: Number of Participants With CHRONIC GVHD
Description: Chronic GVHD is graded by NIH guidelines for chronic GVHD, which evaluates skin, joints, oral, ocular, hepatic, esophagus, GI, respiratory, platelet, and musculoskeletal involvement, in stages from 0 to 3 where 0 means no chronic GVHD, and 3 is the highest stage of chronic GVHD.
Time Frame: Assessed monthly from month 3 to month 12
Population: The analysis included all participants who underwent allogeneic hematopoietic stem cell transplantation (SCT) and were evaluable for chronic GVHD. A participant is evaluable for chronic GVHD if he/she engrafted and survived or remained in the study for more than 100 days after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 8
Participants | 1

9. Primary Outcome: Event-free Survival
Description: Event-free survival is calculated from the date of transplant to the date of graft failure, disease recurrence or death from any cause.
Time Frame: up to 2 years post transplant
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probability of event-free survival
Arm/Group | Bone Marrow or Stem Cell Infusion
Number analyzed (Participants) | 10
probability of event-free survival | 0.7 [0.33 to 0.89]

ADVERSE EVENTS:
Time Frame: Primary BMT studies have a critical toxicity period of 30 days after BMT day 0. During the critical toxicity period the most severe grade of all AE's is captured. Grade 1 and 2 AEs, hematological toxicities, and fevers are excluded. Serious Adverse Events/Unanticipated Problems are reported (excluding hematological toxicities and fevers) until 100 days after BMT day 0.
Description: All adverse events were collected using CTCAE 2.0 for the study. For reporting purpose, adverse event terms were converted using CTCAE v4.0.
Arm/Group | Bone Marrow or Stem Cell Infusion
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow or Stem Cell Infusion (N=10)
Catheter related Infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow or Stem Cell Infusion (N=10)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (6)
Cardiac disorders-Other: Cardiomegaly (Cardiac disorders) | 1 (1)
Catheter Related Infection (Infections and infestations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dysuria (painful urination) (Renal and urinary disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
GGT increased (Investigations) | 5 (20)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hepatobiliary disorders-Other: GVHD (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders-Other: hepatic VOD (Hepatobiliary disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (30)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infections and infestations - Other: Parainfluenza virus (Infections and infestations) | 1 (1)
Infections and infestations - Other: CMV reactivation (Infections and infestations) | 1 (1)
Infections and infestations - Other: Gram negative rods (Infections and infestations) | 2 (3)
Infections and infestations - Other: BK virus (Infections and infestations) | 3 (4)
Infections and infestations - Other: HSV (Infections and infestations) | 1 (1)
Lipase (Investigations) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Nervous system disorders-Other: Altered mental status (Nervous system disorders) | 1 (1)
Eye disorders -Other: PRES (Eye disorders) | 1 (1)
Pain (General disorders) | 1 (3)
Partial thromboplastin time (PTT) (Investigations) | 1 (1)
Pelvic Pain (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (10)
Prothrombin time (PT) (Investigations) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders-Other: Nitrite in urine (Renal and urinary disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (31)
Alanine aminotransferase increased (Investigations) | 6 (31)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Stomatitis/Pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Wound-Infectious (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes